CLINICAL TRIAL: NCT06716190
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Doses of BI 3731579 in Healthy Volunteers (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Different Doses of BI 3731579 Are Tolerated by Healthy People
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1519-0002; 2024-517209-95-00 (Registry Identifier: CTIS (EU)); U1111-1313-5393 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MRD: BI 3731579 dose group 1 (Experimental): MRD= Multiple rising doses
  Interventions: Drug: BI 3731579; Drug: Midazolam
- MRD: BI 3731579 dose group 2 (Experimental)
  Interventions: Drug: BI 3731579; Drug: Midazolam
- MRD: BI 3731579 dose group 3 (Experimental)
  Interventions: Drug: BI 3731579; Drug: Midazolam
- MRD: BI 3731579 dose group 4 (Experimental)
  Interventions: Drug: BI 3731579; Drug: Midazolam
- MRD: Placebo matching BI 3731579 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3731579; Drug: Midazolam

INTERVENTIONS:
Drug: BI 3731579 — BI 3731579
  Arms: MRD: BI 3731579 dose group 1; MRD: BI 3731579 dose group 2; MRD: BI 3731579 dose group 3; MRD: BI 3731579 dose group 4
Drug: Placebo matching BI 3731579 — Placebo matching BI 3731579
  Arms: MRD: Placebo matching BI 3731579
Drug: Midazolam — Midazolam

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics and pharmacodynamics of BI 3731579 in healthy volunteers following administration of multiple rising doses per day over 15 days.

ELIGIBILITY:
Inclusion criteria

1. Healthy volunteers according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR) and temperature), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion criteria

1. Any finding in the medical examination (including BP, PR, RR, temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or resting pulse rate outside the range of 45 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to Day 27.

SECONDARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of BI 3731579 in plasma at steady state over a uniform dosing interval τ) | up to Day 19.
Cmax,ss (maximum measured concentration of BI 3731579 in plasma at steady state over a uniform dosing interval τ) | up to Day 19.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com